CLINICAL TRIAL: NCT01485887
Title: A Open-label Long-term Extension Study To Evaluate The Safety And Efficacy Of Venlafaxine Er In Adult Outpatients With Major Depressive Disorder
Brief Title: Venlafaxine ER Long-Term Extension Study for Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2411264
Record Dates: First submitted 2011-11-29; First posted 2011-12-06 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder
Keywords: Venlafaxine ER; long-term extension; Japan
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venlafaxine ER (Experimental)
  Interventions: Drug: Venlafaxine ER

INTERVENTIONS:
Drug: Venlafaxine ER — Treatment phase: 10 months (75-225 mg/day), oral administration Tapering phase: 1-3 weeks (stepwise dose reduction: 150-37.5 mg/day), oral administration

SUMMARY:
This is a phase 3, flexible-dose, open-label, multi-center study. The subjects who complete the week 8 visit in the prior double-blind study (B2411263) will be eligible to participate in this study. This study consists of 10 month treatment phase and 1-3 week tapering phase. The 2 follow-up visits will be evaluated after 2 weeks and 4 weeks of last study medication dosing.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed 8 weeks double-blind study (B2411263), without major protocol violations or tolerability concerns in the opinion of the investigator.

Exclusion Criteria:

* Clinically important abnormalities on baseline (Week 8 of the double-blind study) physical examination, or any unresolved clinically significant abnormalities on electrocardiogram (ECG), laboratory test results, or vital signs recorded before Week 8 in the previous double-blind study.
* Significant risk of suicide based on clinical judgment.
* Use of prohibited treatments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- Japan (25):
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai, Chiba
  - Nakamoto Clinic, Noda, Chiba
  - Stress Care Yoshimura Clinic, Fukuoka, Fukuoka
  - Hatakeyama Clinic, Kitakyushu, Fukuoka
  - Shiranui Hospital, Omuta, Fukuoka
  - Fujikawa Clinic, Hatsukaichi, Hiroshima
  - Takahashi Psychiatric Clinic, Ashiya, Hyōgo
  - Ikeuchi Psycho Induced Internal Med.Clinic, Kobe, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Medical Corporation Seishinkai Kishiro Mental Clinic, Kawasaki, Kanagawa
  - Yutaka Clinic, Sagamihara-shi, Kanagawa
  - Tawara Clinic, Yokohama, Kanagawa
  - Shioiri Mental Clinic, Yokosuka, Kanagawa
  - Shibamoto Clinic, Osakasayama-shi, Osaka
  - Suzuki Hospital, Adachi-ku, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Setagaya-ku, Tokyo
  - Omotesando Mental Clinic, Shibuya-ku, Tokyo
  - Maynds Tower Mental Clinic, Shibuya-ku, Tokyo
  - Tokyo Kosei Nenkin Hospital, Shinjuku-ku, Tokyo
  - Himorogi Psychiatric Institute, Toshima-ku, Tokyo
  - Tenjin Mental Clinic, Fukuoka
  - Stress Care Yoshimura Clinic, Fukuoka
  - Kuranari Psychiatry Clinic, Fukuoka
  - Medical Corporation Toyokokai Tawara Clinic, Kanagawa
  - Sagaarashiyama-Tanaka Clinic, Kyoto

REFERENCES:
- [Derived] Higuchi T, Kamijima K, Nakagome K, Itamura R, Asami Y, Kuribayashi K, Imaeda T. A randomized, double-blinded, placebo-controlled study to evaluate the efficacy and safety of venlafaxine extended release and a long-term extension study for patients with major depressive disorder in Japan. Int Clin Psychopharmacol. 2016 Jan;31(1):8-19. doi: 10.1097/YIC.0000000000000105. PMID 26513202
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2411264&StudyName=Venlafaxine%20ER%20Long-Term%20Extension%20Study%20for%20Major%20Depressive%20Disorder%20%28MDD%29

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who have completed the week 8 visit in the preceding double-blind study B2411263 (NCT01441440) were eligible to participate in this study.
Groups:
- Venlafaxine ER 75-225 mg/Day Flexible: Participants orally received venlafaxine ER once daily after dinner or breakfast at a dosage within the predetermined range (75, 150, and 225 mg/day). Participants commenced venlafaxine ER treatment at the dosage of 37.5 mg/day, and after 1 week, increased the dosage to 75 mg/day and continued treatment for 1 week. If no tolerability issue was observed after 2 weeks by the judgment of the investigators, the dosage was increased to 150 mg/day and continued for 1 week. Furthermore, if no tolerability issue was observed after 3 weeks by the judgment of the investigators, the dosage was increased to 225 mg/day. Participants were able to remain at the same dose by the judgment of investigators if there was any tolerability concern from dose escalation. In addition, dose reduction was allowed upon occurrence of tolerability concern following dose escalation.
Period: Overall Study
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Started | 50
Completed | 38
Not Completed | 12
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 8
Not completed — Deterioration of primary disease | 1
Not completed — Primary disease markedly improved | 1

BASELINE CHARACTERISTICS:
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 26
  MALE | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an adverse event (AE), without regard to possibility of causal relationship. Treatment-emergent adverse events: those which occurred or worsened after baseline. An AE resulting in any of the following outcomes, was considered to be a serious adverse event: death; lifethreatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]) up to 10 months
Population: Participants who recieved at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Participants
  Adverse events (AEs) | 49
  Serious adverse events (SAEs) | 2

2. Primary Outcome: Number of Participants With Clinical Significant Vital Changes
Description: Clinical significant changes were pre-defined for systolic blood pressure (SBP), diastolic blood pressure (DBP) , and pulse rate (PR). An average value of 3 measurements in each visit meeting the following criteria for 3 consecutive visits was determined as clinical siginificant changes: DBP >= 90 mmHg with change from the baseline >= 10 mmHg; SBP >= 140 mmHg with change from the baseline >= 20 mmHg; PR >= 100 bpm with change from the baseline >= 15 bpm.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]) up to 10 months
Population: Participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Participants
  Systoloc blood pressure (SBP) | 3
  Diastolic bloodpressure (DBP) | 4
  Pulse rate | 1

3. Primary Outcome: Number of Participants With Clinical Significant Laboratory Tests Changes
Description: Clinical significant changes were pre-defined for each laboratory test based on the criteria: Red Blood Cell Count <0.8 x lower limit normal (LLN); Lymphocytes (%) <0.8 x LLN; Eosinophils (%) >1.2 x upper limit normal (ULN); Total Bilirubin >1.5 x ULN; Alanine Aminotransferase (ALT) >3.0 x ULN; Gamma glutamyl transferase (GGT) >3.0 x ULN; Uric Acid >1.2 x ULN; Cholesterol >1.3 x ULN; Low density lipoprotein (LDL) cholesterol >1.2 x ULN; Triglycerides >1.3 x ULN; Glucose >1.5 x ULN; Urine Glucose [qualitative (Qual)] >=1; Urine Protein (Qual) >=1; Urine Blood/Hemoglobin (Hgb) (Qual) >=1.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]) up to 10 months
Population: Participants with at least one observation of the given laboratory test while on study treatment or during lag time.
Measure: Number; unit: Participants
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 49
Participants
  Red Blood Cell Count < 0.8xLLN | 1
  Lymphocytes (%) < 0.8xLLN | 2
  Eosinophils (%) > 1.2xULN | 3
  Total Bilirubin > 1.5xULN | 1
  ALT > 3.0xULN | 1
  GGT > 3.0xULN | 4
  Uric Acid > 1.2xULN | 1
  Cholesterol > 1.3xULN | 4
  LDL Cholestero l> 1.2xULN | 12
  Triglycerides > 1.3xULN | 8
  Glucose > 1.5xULN | 3
  Urine Glucose (Qual) >= 1 | 3
  Urine Protein (Qual) >= 1 | 3
  Urine Blood/Hgb(Qual) >= 1 | 10

4. Primary Outcome: Number of Participants With Clinical Significant Electrocardiogram (ECG) Changes
Description: Clinically significant ECG findings included: corrected QT (QTc), QT interval corrected using the Bazett's formula (QTcB), and QT interval corrected using the Fridericia formula (QTcF)> 450 millisecond (ms), >480 ms, and >500 ms respsctively, change from baseline in QTc, QTcB, and QTcF >= 30 ms, and >= 60 ms, respectively.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]) up to 10 months
Population: Participants with at least one observation of the electrocardiogram while on study treatment.
Measure: Number; unit: Participants
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 49
Participants
  QT Interval > 450 ms | 5
  QT Interval > 480 ms | 0
  QT Interval > 500 ms | 0
  QTcB Interval > 450 ms | 17
  QTcB Interval > 480 ms | 4
  QTcB Interval > 500 ms | 1
  QTcF Interval > 450 ms | 8
  QTcF Interval > 480 ms | 1
  QTcF Interval > 500 ms | 0
  QT Interval increase from baseline >= 30 ms | 7
  QT Interval increase from baseline >= 60 ms | 0
  QTcB Interval increase from baseline >= 30 ms | 8
  QTcB Interval increase from baseline >= 60 ms | 0
  QTcF Interval increase from baseline >= 30 ms | 4
  QTcF Interval increase from baseline >= 60 ms | 0

5. Primary Outcome: Number of Participants With no at Baseline and Yes at Any Post Baseline for Columbia Suicide-Severity Rating Scale (C-SSRS) According to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories
Description: C-SSRS is a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Yes/No responses are mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories: Completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. A participant could have a yes or no response in more than one category.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]) up to 10 months
Population: Participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Participants
  Completed suicide | 0
  Suicide attempt | 0
  Preparatory acts toward imminent suicidal behavior | 0
  Suicide ideation | 0
  Self-injurious behavior, no suicidal intent | 0

6. Secondary Outcome: Change From Baseline in 17-item Hamilton Rating Scale for Depression (HAM-D17) at Each Post Baseline Time Point
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression (symptoms such as depressed mood, work and activities, sleep, suicide, psychomotor agitation/retardation, appetite, sexual interest, anxiety, and somatic symptoms). The items of the HAM-D17 are rated on a scale of 0 to 2 (8 items) or 0 to 4 (9 items), and the total score ranges from 0 to 52. Higher scores indicate more severe symptoms. Change from baseline: mean score at observation minus mean score at baseline.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]), Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44
Population: Participants who recieved at least one dose of study drug in this study , and had at least one evaluable HAM-D17 score after Week 8 of the preceding study B2411263 (NCT01441440). 'n' is signifying those participants who were evaluated for this measure at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Units on a scale
  Week 1 (n=50) | -1.0 (2.00)
  Week 2 (n=50) | -1.5 (3.47)
  Week 3 (n=50) | -2.2 (4.76)
  Week 4 (n=50) | -2.9 (4.55)
  Week 6 (n=47) | -3.4 (4.39)
  Week 8 (n=48) | -3.9 (4.61)
  Week 12 (n=47) | -4.1 (5.41)
  Week 16 (n=46) | -4.4 (7.06)
  Week 20 (n=45) | -6.2 (4.93)
  Week 24 (n=44) | -5.7 (5.08)
  Week 28 (n=42) | -6.1 (5.67)
  Week 32 (n=41) | -6.4 (5.81)
  Week 36 (n=41) | -6.5 (5.85)
  Week 40 (n=40) | -6.4 (6.55)
  Week 44 (n=40) | -7.1 (5.98)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) at Each Post Baseline Time Point
Description: CGI-S is a 7-point clinician rated scale to assess severity of participant's current illness state; range: 1=normal, not ill at all, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill patients. Higher scores reflect higher severity of current illness states. Change from baseline: mean score at observation minus mean score at baseline.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Units on a scale
  Week 1 (n=50) | -0.1 (0.46)
  Week 2 (n=50) | -0.3 (0.63)
  Week 3 (n=50) | -0.3 (0.87)
  Week 4 (n=50) | -0.4 (0.81)
  Week 6 (n=47) | -0.6 (0.77)
  Week 8 (n=48) | -0.6 (0.91)
  Week 12 (n=47) | -0.8 (1.20)
  Week 16 (n=46) | -0.9 (1.34)
  Week 20 (n=45) | -1.2 (0.98)
  Week 24 (n=44) | -1.1 (1.01)
  Week 28 (n=42) | -1.2 (1.07)
  Week 32 (n=41) | -1.2 (1.11)
  Week 36 (n=41) | -1.2 (1.19)
  Week 40 (n=40) | -1.2 (1.23)
  Week 44 (n=40) | -1.3 (1.12)

8. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Score at Each Post Baseline Time Point
Description: CGI-I is a 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Scores above 4 reflect worsening of illness state as compared to baseline.
Time Frame: Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 50
Units on a scale
  Week 1 (n=50) | 3.8 (0.62)
  Week 2 (n=50) | 3.5 (0.81)
  Week 3 (n=50) | 3.3 (1.05)
  Week 4 (n=50) | 3.1 (1.05)
  Week 6 (n=47) | 2.9 (0.91)
  Week 8 (n=48) | 2.9 (0.96)
  Week 12 (n=47) | 2.6 (1.06)
  Week 16 (n=46) | 2.4 (1.20)
  Week 20 (n=45) | 2.1 (0.97)
  Week 24 (n=44) | 2.2 (1.05)
  Week 28 (n=42) | 2.2 (1.09)
  Week 32 (n=41) | 2.1 (1.14)
  Week 36 (n=41) | 2.2 (1.18)
  Week 40 (n=40) | 2.1 (1.25)
  Week 44 (n=40) | 2.0 (1.15)

9. Secondary Outcome: Change From Baseline in 16-item Quick Inventory of Depressive Symptomatology Self-Report Japanese Version (QIDS16-SR-J) at Each Post Baseline Time Point
Description: QIDS16-SR-J is a self-rated scale used in patients with major depressive disorder to measure the overall severity of depressive symptoms: 1) sad mood; 2) concentration; 3) self-criticism; 4) suicidal ideation; 5) interest; 6) energy/fatigue; 7) sleep disturbance (initial, middle, and late insomnia or hypersomnia); 8) decrease/increase in appetite/weight; and 9) psychomotor agitation/retardation. QIDS16-SR-J items are rated on a scale of 0 to 3, and the total score ranges from 0 to 27. Higher scores indicate more severe symptoms. Change from baseline: mean score at observation minus mean score at baseline.
Time Frame: Baseline (Week 8 of the preceding double-blind study B2411263 [NCT01441440]), Weeks 12, 24, 44
Population: Participants who recieved at least one dose of study drug in this study , and had at least one evaluable HAM-D17 score and QIDS16-SR-J score after Week 8 of the preceding study B2411263 (NCT01441440). 'n' is signifying those participants who were evaluated for this measure at each time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Number analyzed (Participants) | 49
Units on a scale
  Week 12 (n=47) | -2.7 (4.97)
  Week 24 (n=44) | -3.8 (4.45)
  Week 44 (n=40) | -4.7 (4.73)

ADVERSE EVENTS:
Arm/Group | Venlafaxine ER 75-225 mg/Day Flexible
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine ER 75-225 mg/Day Flexible (N=50)
Pyrexia (General disorders) | 1
Crime (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine ER 75-225 mg/Day Flexible (N=50)
Palpitations (Cardiac disorders) | 5
Hyperacusis (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 4
Vertigo (Ear and labyrinth disorders) | 2
Blepharospasm (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 2
Fatigue (General disorders) | 1
Feeling abnormal (General disorders) | 6
Irritability (General disorders) | 2
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Thirst (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 3
Seasonal allergy (Immune system disorders) | 3
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 20
Sinusitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Overdose (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 2
Blood pressure increased (Investigations) | 7
Electrocardiogram QT prolonged (Investigations) | 2
Electrocardiogram T wave inversion (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Heart rate increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Occult blood positive (Investigations) | 1
Protein urine present (Investigations) | 1
Weight decreased (Investigations) | 3
Weight increased (Investigations) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperphagia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 13
Hyperaesthesia (Nervous system disorders) | 1
Hypersomnia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Retrograde amnesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 9
Tethered cord syndrome (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Acute stress disorder (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Initial insomnia (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Loss of libido (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.